CLINICAL TRIAL: NCT01757392
Title: Study of the Safety and Effectiveness of Candin for the Treatment of Common Warts
Brief Title: Candin Safety & Efficacy Study for the Treatment of Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nielsen BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nieslen Protocol CFW-2c
Record Dates: First submitted 2012-12-21; First posted 2012-12-28 (Estimated); Results first posted 2021-01-11 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Warts; Human Papilloma Virus
Keywords: Treatment; common wart lesions; (verruca vulgaris)
MeSH Terms: conditions — Warts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Candin® 0.3 mL (Experimental): Monthly intralesional injections of Candin® 0.3 ml until lesion resolves or up to 6 injections.
  Interventions: Biological: Candida albicans Skin Test Antigen

INTERVENTIONS:
Biological: Candida albicans Skin Test Antigen — 0.3 ml injected intralesionally monthly. Number of injections: until wart lesion is resolved or up to 6 injections.
  Other Names: Candin®

SUMMARY:
The primary objective of this study is to determine the safety of Candin® (Candida albicans Skin Test Antigen) at a 0.3 ml dose level at up to 6 monthly injections for treating common warts (Verruca vulgaris).

DETAILED DESCRIPTION:
The primary objective of this study is to determine the safety of Candin® (Candida albicans Skin Test Antigen) at either 0.3 mL dose levels at up to 6 monthly injections (a maximal, cumulative dose of 1.9 mL, including the delayed-type hypersensitivity (DTH) test) for treating common warts (Verruca vulgaris). A secondary objective is to understand the relative effectiveness of the 0.3 dose level for treating common warts, both those that were injected and those that were not injected as well as other types of warts that were not injected to allow a determination of appropriate dose levels to use in a future dose-ranging efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 3 and not more than 10 common warts not located on the palms or digits
* Positive DTH response to Candin® required

Exclusion Criteria:

* No previous medical treatment for warts other than OTC
* No immunocompromising medical conditions or medicines allowed
* No preexisting inflammatory conditions at treatment site allowed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandy M Johnson, MD, Principal Investigator — Johnson Dermatology
Locations (1):
- Johnson Dermatology, Fort Smith, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Candin® 0.3 mL: Monthly intralesional injections of Candida albicans Skin Test Antigen 0.3 ml into single wart until lesions resolve or up to 6 injections.
Period: Overall Study
Arm/Group | Candin® 0.3 mL
Started (Number of participants who were screened) | 39
Completed (Number of participants who received at least one wart injection) | 35
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Screen Fail | 3

BASELINE CHARACTERISTICS:
Population: ITT population/ Safety Population
Groups:
- Candin® 0.3 mL: Monthly intralesional injections of Candida albicans Skin Test Antigen 0.3 ml into single wart until lesion resolves or up to 6 injections.
Arm/Group | Candin® 0.3 mL
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 34
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 35
Weight [Mean (Standard Deviation); unit: Kg] | 87.32 (22.508)
Height [Mean (Standard Deviation); unit: cm] | 173.52 (10.982)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.66 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Resolution of Primary Injected Wart
Time Frame: Monthly evaluations during injection visit for up to 5 months, the follow up visits at 1 and 4 months after last dose for a total of approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Candin® 0.3 mL
Number analyzed (Participants) | 35
Participants | 19

2. Secondary Outcome: Number of Participants With Complete Resolution of the Primary Injected Wart by Number of Injection Visits
Time Frame: as for outcome 1
Population: Subjects experiencing complete resolution of the primary injected wart
Measure: Count of Participants; unit: Participants
Arm/Group | Candin® 0.3 mL
Number analyzed (Participants) | 19
Participants
  One Injection visit | 5
  Two Injection visits | 4
  Three Injection visits | 3
  Four Injection visits | 4
  Five Injection visits | 1
  Six Injection visits | 2

3. Post Hoc Outcome: Number of Participants With Complete Resolution of the First Non-injected Wart by Injection Visits
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Candin® 0.3 mL
Number analyzed (Participants) | 18
Participants
  One injection visit | 5
  Two injection visits | 2
  Three Injection visits | 5
  Four Injection visits | 1
  Five Injection visits | 0
  Six Injection visits | 5

4. Post Hoc Outcome: Number of Participants With Complete Resolution of All Qualified Warts by Injection Visits
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Candin® 0.3 mL
Number analyzed (Participants) | 12
Participants
  One injection visit | 0
  Two injection visits | 0
  Three injection visits | 2
  Four injection visits | 4
  Five injection visits | 3
  Six injection visits | 3

5. Post Hoc Outcome: Recurrence of Resolved Primary Wart at Follow up 2 Visit
Description: Number of participants with recurrence of primary wart seen at the final follow up visit
Time Frame: 4 months after last injection
Measure: Count of Participants; unit: Participants
Arm/Group | Candin® 0.3 mL
Number analyzed (Participants) | 19
Participants | 4

ADVERSE EVENTS:
Time Frame: All Post Dose visits over approximately 9 months, including treatment phase (5 months) and follow up period (4 months)
Groups:
- Candin® 0.3 mL: Monthly intralesional injections of Candida albicans Skin Test Antigen 0.3 ml until lesion resolves or up to 6 injections.
Arm/Group | Candin® 0.3 mL
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 1/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Candin® 0.3 mL (N=35)
Cholecystitis (Hepatobiliary disorders) | 1 (1) — cholecystitis followed by cholecystectomy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candin® 0.3 mL (N=35)
Injection site erythema (General disorders) | 32
Injection site Pain (General disorders) | 32
Injection site swelling (General disorders) | 31
Injection site pruritus (General disorders) | 20
Headache (Nervous system disorders) | 11
Fatigue (General disorders) | 10
Injection site exfoliation (General disorders) | 9
Influenza like illness (General disorders) | 8
Diarrhea (Gastrointestinal disorders) | 5
Injection site vesicles (General disorders) | 5
Nausea (Gastrointestinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 2
Alanine aminotranferase increased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes